CLINICAL TRIAL: NCT04737408
Title: Influence of Intensive Lipid-lowering With Statin and Ezetimib Prescription on Computed Tomography Derived Fractional Flow Reserve in Patients With Stable Chest Pain (The FLOW-PROMOTE Study)
Brief Title: Influence of Intensive Lipid-lowering on FFRCT (The FLOW-PROMOTE Study)
Acronym: FlowPromote
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bjarne Linde Noergaard (Other)
Responsible Party: Sponsor-Investigator, Bjarne Linde Noergaard, Associate Professor, MD, PhD, FESC, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Aarhus University Hospital
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease, fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Intervention Model Description: Patients are randomized 1:1 to two different lipid lowering medical treatment strategies
Masking Description: Open label design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Usual care" (Active Comparator): "Usual care" prevention: atorvastatin 40 mg per day for 18 months
  Interventions: Drug: Rosuvastatin 40mg
- "Intensive care" (Experimental): "Intensive care" prevention: rosuvastatin 40 mg + ezetimib 10 mg per day for 18 months
  Interventions: Drug: Rosuvastatin 40mg

INTERVENTIONS:
Drug: Rosuvastatin 40mg — Rosuvastatin 40 mg
  Other Names: Ezetimib 10mg

SUMMARY:
The FLOW-PROMOTE Study is an investigator-initiated, Danish multicenter study of patients with stable chest pain investigating whether lipid lowering is associated with recovery of impaired coronary flow as assessed by CT derived fractional flow reserve (FFRCT).

DETAILED DESCRIPTION:
Multicenter study (4 centers in Denmark), including 120 patients with stable chest pain and hemodynamically significant coronary artery disease as assessed by FFRCT. By using two lipid lowering treatment strategies ("usual" vs "intensive" care) over 18 months, the effect on coronary plaque regression and flow recovery are assessed from repeated CT angiograms with plaque and FFRCT analyses at 9 and 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms suggestive of stable coronary artery disease (CAD)
2. No known CAD
3. At least one coronary stenosis with >49% lumen reduction determined by CT angiography
4. Sinus rhythm
5. At least one lesion with FFRCT <0.81 (see below)
6. Life expectancy >3 years
7. Fertile women must use safe contraception throughout the study period
8. Signed informed consent

5. LDL cholesterol >2.0 mM (patients already on lipid lowering medical therapy < 3 months can be included if meeting all of the above mentioned criteria)

Exclusion Criteria:

1. Unstable angina
2. Known CAD
3. Body mass index >40
4. Allergy to iodinated contrast media
5. Known statin intolerance
6. Poor coronary CT angiography image quality inadequate for FFRCT calculation (determined by core-laboratory)
7. Significant left main coronary artery (stenosis >49%) or three-vessel CAD determined by coronary CT angiography leading to direct referral to ICA
8. FFRCT <0.81 over the left main coronary artery or the proximal left anterior descendens artery (LAD) segment, or <0.76 over the mid-LAD, proximal circumflex, right coronary artery or intermediate coronary segments
9. Pregnancy (women with age >45 will be screened for pregnancy)
10. Moderate to severe liver failure
11. Estimated glomerular filtration rate (eGFR) < 60 ml/min
12. Participation in another trial
13. Does noes not wish to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
18-month change in coronary flow | 18 months
  Coronary flow will be assessed by repetitive FFRCT assessments (0,9 and 18 months)

SECONDARY OUTCOMES:
18-month change high risk coronary plaque volumes | 18 months
  Will be assessed by measuring low attenuation coronary plaque (LAP) volumes at repetitive CT angiograms (0,9, and 18 months)
18-month change in high risk coronary plaque features | 18-months
  Will be assessed by quantifying the proportion of lesions with positive remodeling at repetitive CT angiograms (0,9, and 18 months).
18-month change in coronary vessel volumes | 18-months
  Will be assessed by calculating the vessel volume relative to myocardial mass (V/M) ratio determined from repetitive CT angiograms (0,9, and 18 months).
18-month change in indices of coronary inflammation | 18-months
  Will be assessed by the pericoronary fat attenuation index (FAI) determined from repetitive CT angiograms (0,9, and 18 months).

OTHER OUTCOMES:
Reproducibility assessment | 9-months
  There will be performed 2 CTA investigations at the 9 month follow-up. Reproducibility assessment of CT derived FFR, plaque markers, FAI and V/M ratio will be performed by calculation of standard error of measurement and within-subject coefficient of variation.

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne L Noergaard, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Southwestern Hospital Esbjerg, Esbjerg
  - Lillebaelt Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No